CLINICAL TRIAL: NCT01608529
Title: Phase 1: Effects of a Restriction Device Ventilatory Nasal Flow on Pulmonary Ventilation and Gas Exchange During Exercise
Brief Title: Feel Breathe, Restriction Device Ventilatory Nasal
Acronym: FB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Cadiz (Other)
Collaborators: Consejo Superior de Deportes, Spain (Other); European Regional Development Fund (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC26392
Record Dates: First submitted 2012-05-17; First posted 2012-05-31 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Mouth Breathing; Restrictive Breathing Pattern
Keywords: Restriction device ventilatory nasal flow; oronasal breathing; nasal breathing.
MeSH Terms: conditions — Mouth Breathing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cyclist group (Experimental)
  Interventions: Device: Feel Breathe, restriction device ventilatory nasal

INTERVENTIONS:
Device: Feel Breathe, restriction device ventilatory nasal — The Feel Breathe (FB) consisted of a small adhesive strip that is placed across the bridge of the nose during exercise. The FB was place following procedures for placement as indicated by the manufacturer's directions, while the placebo nasal, was placed over the nostrils of the subject, without interfering nasal breathing; thus, nasal airflow resistance was not increase. Each subject was required to perform three identical submaximal exercises with intensity at 50% VT1-VT2 under different breathing conditions. The breathing conditions were: oronasal, nasal and FB breathing. All participants performed three trials of stable load (50% VT1-VT2) for 10 minutes in the three conditions mentioned above, setting the cadence at 70-75 rpm, and controlling the same in all three exercise conditions.
  Other Names: Restriction device ventilatory nasal. PCT/ES2010/000429.; Feel Breathe. Registro: N0299875-0.

SUMMARY:
It has patented a restriction and filtering device ventilatory nasal flow FeelBreathe with the aim of increase nasal airflow resistance, therefore the objective was to examine the effects of FeelBreathe with lung ventilation and gas exchange during exercise.

DETAILED DESCRIPTION:
Background: Different devices are currently used to train inspiratory muscles, thus showing an increase in the physical performance. It is a control trial to investigate the effects of a new restriction and filtering device ventilatory nasal flow (FeelBreathe).

Methods: A total of 27 trained male caucasian subjects (age: 32.5 ± 7.23 years) were recruited from different sports clubs. Measurement of maximum static inspiratory pressure were taken before exercise testing and an incremental test in cycle ergometer to volitional fatigue for the determination of gas exchange data. Each subject performed three identical submaximal exercises at 50% of ventilatory thresholds under different breathing conditions: 1) oronasal breathing 2) nasal breathing and 3) nasal breathing with Feel Breathe, Restriction and Filtering Device Ventilatory Nasal Flow.

Discussion: Researchers try to find if the new device called FeelBreathe causes changes in the lung ventilation and gas exchange during exercise. If the results show altered breathing pattern and cardiometabolic variables, FeelBreathe could be used to training respiratory muscles.

ELIGIBILITY:
Inclusion Criteria:

* Age: 25-35 years.
* trained male caucasian cyclists
* Non-smokers
* Each subject completed an approved informed consent form and detailed health questionnaire before testing.

Exclusion Criteria:

* Smokers.
* Presence of diseases during the test period. In particular, they had no current symptoms of nasal disease, snoring, asthma or allergic rhinitis.
* Unwillingness to complete the study requirements.

Ages: 25 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Overall Impact of a restriction device ventilatory nasal over different physiological variables in cyclists | Subjects were assessed during 8 weeks
  VE (l/min), Vtin (ml/kg), BF (bf/min), VCO2 (ml/min), VE/VO2 (ml), VE/VCO2 (ml), RER (VCO2/VO2), PETO2 (mmHg), PETCO2 (mmHg), tin (s/insp), tex (s/expir), Vtin (ml/min), Vtex (ml/min), SPO2 (%) and VO2 (ml/kg/min) were assessed throughout the exercise on a cycle ergometer (ERGO-Line GmbH + CoKG, mod. Jaeger ER-900. Germany) using three different conditions of breathing: oronasal, nasal and nasal breathing with FeelBreathe, with 10-sec sampling intervals using a open circuit spirometry (CPX Cardinal Health, 234 GmbH, Leibnizstrasse 7, D-97204 Hoechberg, Germany).

SECONDARY OUTCOMES:
Maximum oxygen uptake | Subjects were assessed during 8 weeks
  Before experimental trials each subject performed a incremental protocol on a cycle ergometer (ERGO-Line GmbH + CoKG, mod. Jaeger ER-900. Alemania) for the determination of gas exchange. The test was stopped upon volitional fatigue of the subject gas-exchange data were measured breath-by-breath using open circuit spirometry (CPX Cardinal Health, 234 GmbH, Leibnizstrasse 7, D-97204 Hoechberg, Alemania).
Maximum static inspiratory pressure (PImax) | Subjects were assessed during 8 weeks
  Inspiratory muscle testing was performed using a mouth pressure meter (Micro Medical Inc., Chatham, Kent, UK). The manufacturer states that the test-retest reliability of this device is ±3%. Maximum static inspiratory pressure was measured at residual volume and the best result from three inspiratory attempts was taken. At least one minute was allowed between attempts to minimize the effects of muscle fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Lopez Chicharro, MD, Principal Investigator — Universidad Complutense de Madrid; Jorge dR Fernandez Santos, Phd Student, Study Chair — University of Cádiz (Spain); Davinia Vicente Campos, Phd, Study Chair — Universidad Complutense de Madrid; Carmen Vaz Pardal, MD, Study Chair — Centro de Medicina del Deporte (Cádiz); Jose L Costa Sepulveda, Phd Student, Study Chair — University of Cádiz (Spain); Jose L Gonzalez Montesinos, Phd, Study Director — University of Cádiz (Spain); Jose Castro Piñero, Phd, Study Director — University of Cádiz (Spain); Julio Conde Caveda, Phd, Study Director — University of Cádiz (Spain)
Locations (1):
- Centro de Medicina del Deporte, San Fernando, Cadiz, Spain